CLINICAL TRIAL: NCT05773924
Title: Evaluation of Efficacy and Safety of the triLift™ System
Acronym: LUM-triLift
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lumenis Be Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LUM-ABU-triLift-22-01
Record Dates: First submitted 2023-02-23; First posted 2023-03-17 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-02

CONDITIONS: Skin Laxity; Wrinkle
Keywords: laxity, facial lifting, wrinkles, rhytids
MeSH Terms: conditions — Cutis Laxa

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Trilift system treatment arm (Other): Single arm with Before & After photos, triLift treatment protocol study design.
  Interventions: Device: triLift system

INTERVENTIONS:
Device: triLift system — To evaluate the efficacy of the triLift™ treatment

SUMMARY:
Single center, single-arm, prospective, open Label with Before & After Study Design.

DETAILED DESCRIPTION:
Single center, single-arm, prospective, open Label with Before & After Study Design. The control group will be the subjects before the triLift™ treatment protocol and the experimental group will consist of the same subjects after completion of the triLift™ treatment protocol.

ELIGIBILITY:
Inclusion Criteria:

* Subject is willing and able to read, understand, and sign the informed consent.
* Healthy male or female aged 35 - 55 years.
* Fitzpatrick skin type 1-6.
* Subject is capable of reading, understanding, and following instructions of the procedure to be applied.
* Subject is able and willing to comply with the treatment. Women in childbearing age who is willing to conduct a pregnancy test prior to each treatment.

Exclusion Criteria:

* Pregnant, lactating, or plans to become pregnant during the study period or had given birth less than 6 months ago.
* Concurrent participation in any other study.
* Subject has a pacemaker or internal defibrillator, implanted neurostimulators or any other internal electric device or patient who had an implant in the past.
* Subject has metal or other implants in the treatment area (Not including dental fillings, implants and crowns).
* Subject has significant concurrent skin conditions affecting areas to be treated such as sores, bleeding, skin fragility, eczema or psoriasis.
* Subject has burned, blistered, irritated, or sensitive skin due to excessive fresh tanning in areas to be treated or is unlikely to refrain from excessive tanning during the study.
* Subject has used oral isotretinoin (Accutane® or Roaccutan®) within 6 months prior to study.
* Subject has used topical retinoids in the past 1 month.
* History of systemic cancer; premalignant skin lesion or skin concern treatment area.
* Concurrent conditions such as epilepsy, autoimmune, pulmonary or cardiac disorders.
* Poorly controlled endocrine disorders such as diabetes.
* Impaired immune system due to immunosuppressive diseases such as HIV or AIDS, or use of immunosuppressive medications.
* History of collagen disorders, keloid formation or abnormal wound healing.
* Takes or has taken medications, herbal preparations, food supplements or vitamins that might cause fragile skin or impaired skin healing.
* Subject has used oral steroids in the past 6 months.
* Subject has used topical steroids in the past 3 months.
* History of bleeding coagulopathies or use of anticoagulants.
* Use of non-steroidal anti-inflammatory drugs (NSAIDS, e.g. ibuprofen containing agents) one week before and after each treatment session prior to treatment.
* Subjects who cannot feel heat to give proper treatment feedback. (nerve damage, etc.)
* Mental disorders that in the opinion of the Investigator would interfere with the ability to comply with the study requirements.
* Subject has any other medical condition that in the opinion of the Investigator warrants exclusion from this study.

Ages: 35 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-02-10 (Actual); Primary Completion 2023-08-15 (Estimated); Study Completion 2023-08-15 (Estimated)

PRIMARY OUTCOMES:
The Global Aesthetic Improvement scale (GAI) | 4 months
  The Global Aesthetic Improvement scale (GAI) - Success is defined as an improvement of at least 1 point on the GAI scale assessed by the investigator, at the end of the treatment protocol as compared to baseline.

SECONDARY OUTCOMES:
3D images | 4 months
  Measuring facial lifting using 3D imaging and analysis algorithm from Quantificare before and after the treatment protocol
Comfort assessment | 3 months
  Subject assessment of pain and discomfort associated with treatments using a Pain Visual Analogue Scale (VAS), where 0 is "no pain" and 10 is "worst pain possible
Subject level of Satisfaction | 4 months
  Subject satisfaction will be assessed using a 5 level satisfaction questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Arielle Kauvar, MD, Principal Investigator — New York Laser & Skin Care
Locations (1):
- NY Laser Skin Care, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No